CLINICAL TRIAL: NCT01299740
Title: Dialectical Behavioral Therapy (DBT) Based Skills Group for Children With Emotional Dysregulation and Their Parents
Brief Title: Skills Group for Children With Emotional Dysregulation and Their Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Moshe Lachish MD, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR513611CTIL
Record Dates: First submitted 2011-02-13; First posted 2011-02-18 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-02

CONDITIONS: Emotional Dysregulation; Dialectical Behavioral Therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Other): Treatment as usual
  Interventions: Other: Control Group
- Research Group (Experimental): Participation in the DBT skills group
  Interventions: Behavioral: Participation in DBT Skills Group

INTERVENTIONS:
Behavioral: Participation in DBT Skills Group — Participation of 20 group meetings lasting an hour and a half for the children, and 15 group meetings lasting an hour and a half for the parents.
  Arms: Research Group
Other: Control Group — Treatment as usual
  Arms: Control Group

SUMMARY:
Dialectical Behavioral Therapy (DBT) based skill groups for emotionally dysregulated children and their parents

The investigators propose implementing a Dialectical Behavioral Therapy (DBT) skills group format for emotionally dysregulated children between the ages of 8 and 12 and their parents.

Introduction Treatments available for children with emotional dysregulation and behavioral problems were shown to be only partially effective.

DBT combines the western principles of changing behavior with the eastern principles of acceptance and mindfulness.

Efficacy of DBT has been shown across a number of behavioral problems in adults and has been successfully adapted for adolescents. The next logical step is modification for younger children.

The investigators chose DBT because of the observed similarities between adults and adolescents diagnosed with borderline personality disorder and the children who are referred to the investigators clinic with emotional dysregulation.

Aims: To assess the ability to regulate emotions and problem behaviors before and after the proposed intervention

Method:

Population: Between 6-10 children between the ages 8-12 will be recruited from The child and adolescent psychiatric outpatient clinic at Soroka University Medical Center.

Inclusion criteria Children suffering from emotional dysregulation All children and at least one parent speak Hebrew Exclusion criteria

1. Schizophrenia
2. Bipolar disorder
3. Psychosis i.e an overt thought disorder
4. Mental retardation
5. Severe learning disorders
6. Pervasive developmental disorders.
7. Children who have suffered brain injury.

Comparison group: Between 6 and 10 children matched for sex, parents age and education, socioeconomic status that fulfill the same clinical criteria for inclusion in the study as the study group. The comparison group will receive treatment as usual.

Procedure The children will participate in a group skills group over 20 sessions, each session an hour and a half. The parents will participate in a group skills group over 15 sessions, each session an hour and a half. Each group will be lead by two therapists. All the children will be evaluated by board certified child and adolescent psychiatrist and will be diagnosed according to the DSM IV-TR. The parents' the child and a teacher who is familiar with the child will fill in questionnaires before the beginning of the group, at the end of the group process and 6 months after the group ends.

The treatment protocol will be based on Linehan's Skills training manual for treating borderline personality disorder and on modifications made by Miller for adolescents. The groups will be conducted according to a treatment manual which will be written accordingly and modified in order to apply the skills to a younger population. Ancillary treatment ( e.g. pharmacotherapy) will be provided on an as needed basis.

The control group the data will be collected at similar intervals to those in the study group.

Written informed consent will be obtained from the child and a legal guardian.

* ‬
* ‬

ELIGIBILITY:
Inclusion Criteria:

* Children suffering from emotional dysregulation
* All children and at least one parent speak Hebrew

Exclusion Criteria:

1. Schizophrenia
2. Bipolar disorder
3. Psychosis i.e an overt thought disorder
4. Mental retardation
5. Severe learning disorders
6. Pervasive developmental disorders.
7. Children who have suffered brain injury.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in behavioral and emotional functioning | 1 year
  We will assess behavioral and emotional functioning before, at the end and 6 months following the intervention. This will be assessed using the Achenbach questionnaires:(CBCL, TRF). Eight sub-areas will be measured at baseline, at the end of the intervention and six months later. The eight sub-scale symptoms are withdrawn, somatic complaints, anxiety and depression. social problems, thought problems. attention problems. aggressive behavior, and delinquent problems (Externalizing and internalizing).

SECONDARY OUTCOMES:
Improvement in social skills, emotional regulation and concentration | 1 Year
  Social skills will be assessed using The Social Skills Rating System Questionnaire, Emotional regulation with The Difficulties in Emotion Regulation Scale, Hyper-activity and attention with the Conners Rating Scales. The parents Expressed emotions i.e. the intensity of criticism, or over-involvement will be assessed using The Five Minute Speech Sample. Behavioral and emotional functioning of the control group will be assessed using the same measures at the same time intervals. We expect to see a significant improvement on all scales in the research group but not in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Lachish, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel